CLINICAL TRIAL: NCT01807975
Title: Forced Oscillation Versus Spirometry in Diagnosing Post Pulmonary Transplant Bronchiolitis Obliterans Syndrome
Acronym: OSCILLOPOUMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/56
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-05

CONDITIONS: Bronchiolitis Obliterans Syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

ARMS (1):
- post allogreffe patients (Experimental): Functional evaluation of distal airway by forced oscillation technique : relevance earlier diagnostic of pulmonary syndrom of oblitérant bronchiolit in post allogreffe patients
  Interventions: Other: Forced oscillation

INTERVENTIONS:
Other: Forced oscillation

SUMMARY:
A study to evaluate the role of forced oscillation in precocious diagnosis of bronchiolitis obliterans syndrome in patients with pulmonary transplant (time difference in detecting distal airways functional impairment by forced oscillation and the standard technique using spirometry).

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 year-old.
* Patients with cardiopulmonary transplant or bilateral lung transplant.
* Clinically stable patients

Exclusion Criteria:

* Patients already diagnosed with bronchiolitis obliterans.
* Respiratory infection.
* Acute graft rejection.
* Mechanical complications (bronchial dehiscence, pneumothorax, pleural effusion).
* Iatrogenic pneumopathy.
* Inability to perform Respiratory function test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time difference in diagnosing distal airways functional disturbance by forced oscillation and by spirometry (standard methode). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital FOCH, Suresnes, Île-de-France Region, France